CLINICAL TRIAL: NCT05552482
Title: Identification of Factors That Predict Early Haemodialysis Arteriovenous Fistula Failure
Brief Title: Identifying Risk Factors (RF) for Early Haemodialysis Arteriovenous Fistula Failure (eAVFF)
Acronym: eAVFF-RF
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-06Obs-CHRMT
Record Dates: First submitted 2022-09-21; First posted 2022-09-23 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-02

CONDITIONS: Arteriovenous Fistula; Hemodialysis; End Stage Chronic Renal Failure
MeSH Terms: conditions — Arteriovenous Fistula; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with ESRD with early AVF failure: Patients with ESRD who underwent AVF access creation surgery with early AVF failure
  Interventions: Other: Identification of predictive factors
- patients with ESRD without early AVF failure: Patients with ESRD who underwent AVF access creation surgery without early AVF failure
  Interventions: Other: Identification of predictive factors

INTERVENTIONS:
Other: Identification of predictive factors — Evaluation of the following variables : age, sex, body mass index, Diabetes mellitus, vascular disease, hematologic disease, venous thromboembolic disease, antiplatelet or anticoagulant treatments, haemodialysis Catheter Insertion, number of comorbid conditions, Venous diameter, Arterial diameter, AVF type, AVF limb, Anasthesia group

SUMMARY:
Arteriovenous fisutla (AVF) is the vascular access of choice for hemodialysis but has a high early failure (eAVFF) rate. eAVFF can be defined as thrombosis/stenosis and Doppler ultrasound (DUS)-based failure-to-mature parameters such as postoperative blood flow (PostQa) < 500 ml/min, AVF-vein diameter (PostVD) < 5 mm, and AVF-vein depth (PostVDepth) ≥ 6 mm. We explored whether common risk factors for eAVFF could predict these eAVFF parameters and venous distensibility: the latter is largely overlooked as a potential eAVFF parameter.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years)
* Patients who had undergone distal (radioradial and radiocephalic) or proximal arteriovenous fistula (AVF) access creation surgery between 2016 and 2021 at the CHR Metz-Thionville.
* Patients who underwent preoperative and postoperative Doppler ultrasound (DUS) ≤ 4 months after surgery.
* Patients with central venous catheter (CVC) at surgery

Exclusion Criteria:

* Patients using the fistula for intermittent plasmapheresis
* Patients with a radiobasilic AVF or arteriovenous graft

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥ 18 years) who had undergone distal (radioradial and radiocephalic) and proximal arteriovenous fistula (AVF) access creation surgery
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2021-10-05 (Actual); Study Completion 2022-12-21 (Actual)

PRIMARY OUTCOMES:
Identification of the pre/perioperative factors that predict early AVF failure (eAVFF) | up to 3 months after AVF creation
  Comparison of preoperative and intraoperative results according to composite factors of arteriovenous fistula failure: Qa blood flow < 500 ml/min, postoperative venous internal diameter PostVD < 5 mm; complications: presence of stenosis, presence of thrombosis; AVF vein depth (external diameter) (PostVDepth) ≥ 6.
  The following variables were compared between groups: age (years) , sex (Man/Women), body mass index (kg/m2), Comorbidities [Diabetes mellitus (yes/no), obesity (yes/no)], Preoperative hemoglobin (g/dl); locoregional anesthesia (yes/no), Central Venous Catether (CVC) use (yes/no); CVC use on same side as AVF (yes/no); AVF on left side of body (yes/no); Distal AVF location (yes/no); Preop AVF vessel diameter (artery and vein; mm).

SECONDARY OUTCOMES:
Identification of the pre/perioperative factors that predict the early postoperative AVF blood flow (PostQa) | up to 3 months after AVF creation
  Comparison of preoperative and intraoperative results according to AVF blood flow (Qa < 500 ml/min) for the following variables: age (years) , sex (Man/Women), body mass index (kg/m2), Diabetes mellitus (yes/no), vascular disease (yes/no), hematologic disease (yes/no), venous thromboembolic disease (yes/no), antiplatelet or anticoagulant treatments (yes/no), haemodialysis Catheter Insertion (yes/no), the number of comorbid conditions (1, 2, 3 and 4), Venous diameter (mm), Arterial diameter (mm), AVF type (Brachiocephalic/Radiocephalic), AVF limb (left/right), Anasthesia group (local/general)
Identification of the pre/perioperative factors that predict the early postoperative venous internal diameter (PostVD) | up to 3 months after AVF creation
  Comparison of preoperative and intraoperative results according to venous internal diameter (PostVD < 5 mm vs > 5 mm) for the following variables: age (years) , sex (Man/Women), body mass index (BMI: kg/m2), Comorbidities (Diabetes mellitus (yes/no), vascular disease (yes/no), hematologic disease (yes/no), venous thromboembolic disease (yes/no), antiplatelet or anticoagulant treatments (yes/no), haemodialysis Catheter Insertion (yes/no), the number of comorbid conditions (1, 2, 3 and 4), Venous diameter (mm), Arterial diameter (mm), AVF type (Brachiocephalic/Radiocephalic), AVF limb (left/right), Anasthesia group (local/general)
Identification of the pre/perioperative factors that predict the early postoperative AVF stenosis and/or thrombosis | up to 3 months after AVF creation
  Comparison of preoperative and intraoperative results according to stenosis and/or thrombosis (stenosis or thrombosis vs no complications) for the following variables: age (years) , sex (Man/Women), body mass index (kg/m2), Diabetes mellitus (yes/no), vascular disease (yes/no), hematologic disease (yes/no), venous thromboembolic disease (yes/no), antiplatelet or anticoagulant treatments (yes/no), haemodialysis Catheter Insertion (yes/no), the number of comorbid conditions (1, 2, 3 and 4), Venous diameter (mm), Arterial diameter (mm), AVF type (Brachiocephalic/Radiocephalic), AVF limb (left/right), Anasthesia group (local/general)
Identification of the pre/perioperative factors that predict the early postoperative skin to AVF distance | up to 3 months after AVF creation
  Comparison of preoperative and intraoperative results according to skin-AVF distance (< 6 mm vs ≥ 6 mm) for the following variables: age (years) , sex (Man/Women), body mass index (kg/m2), Diabetes mellitus (yes/no), vascular disease (yes/no), hematologic disease (yes/no), venous thromboembolic disease (yes/no), antiplatelet or anticoagulant treatments (yes/no), haemodialysis Catheter Insertion (yes/no), the number of comorbid conditions (1, 2, 3 and 4), Venous diameter (mm), Arterial diameter (mm), AVF type (Brachiocephalic/Radiocephalic), AVF limb (left/right), Anasthesia group (local/general)

CONTACTS AND LOCATIONS:
Overall Officials: Zead TUBAIL, MD, Principal Investigator — CHR Metz Thionville Hopital de Mercy
Locations (1):
- CHR Metz-Thionville/Hopital de Mercy, Metz, France